CLINICAL TRIAL: NCT05326659
Title: Efficacy and Safety of Benvitimod Cream in the Retreatment of Mild to Moderate Psoriasis: Retreatment, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Study
Brief Title: Efficacy and Safety of Benvitimod Cream in the Retreatment of Mild to Moderate Psoriasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Zhonghao Pharmaceutical (Unknown)
Responsible Party: Principal Investigator, Zhang jianzhong, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJ201808BWMD
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Psoriasis
Keywords: Benvitimod Cream; Psoriasis; Retreatment
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benvitimod Cream (Experimental): Benvitimod cream, 1%, applied twice daily for 12 weeks after enrolment.
  Interventions: Drug: Benvitimod Cream
- Placebo (Placebo Comparator): Placebo, applied twice daily for 12 weeks after enrolment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Benvitimod Cream — Benvitimod cream, 1%, applied twice daily for 12 weeks after enrolment.
  Arms: Benvitimod Cream
Drug: Placebo — Placebo, applied twice daily for 12 weeks after enrolment.
  Arms: Placebo

SUMMARY:
This is a retreatment, multicenter, randomized, double-blind, placebo-controlled clinical study to evaluate the safety and efficacy of Benvitimod cream, 1% twice daily for the retreatment of mild to moderate stable psoriasis vulgaris in adults. Approximately 390 participants with mild to moderate stable psoriasis vulgaris will be enrolled and randomly divided into two groups in a 2:1 ratio. They will use either the Benvitimod cream or placebo at the skin with psoriasis vulgaris for 12 weeks.

DETAILED DESCRIPTION:
This is a retreatment, multicenter, randomized, double-blind, placebo-controlled clinical study to evaluate the safety and efficacy of Benvitimod cream, 1% twice daily for the retreatment of mild to moderate stable psoriasis vulgaris in adults. Approximately 390 participants with mild to moderate stable psoriasis vulgaris will be enrolled and randomly divided into two groups in a 2:1 ratio. They will use either the Benvitimod cream or placebo at the skin with psoriasis vulgaris for 12 weeks.

The primary objective is to evaluate the efficacy and safety of Benvitimod cream in the long-term (intermittent) treatment of mild to moderate psoriasis vulgaris. The primary endpoint is proportion of participants with ≥75% improvement in Psoriasis Area and Severity Index (PASI) score 12 weeks after retreatment with Benvitimod cream or placebo.

The study is anticipated to last from April 2022 to August 2023 with 390 participants recruited form about 20 centers in China. All the related investigative organization and individuals will obey the Declaration of Helsinki and Chinese Good Clinical Practice standard. The study has been approved by Institutional Review Board (IRB) and Ethics Committee (EC) in Peking University People's Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age 18~65 years.
* Patients who were treated with Benvitimod cream and have discontinued medication were again diagnosed as suitable for treatment with Benvitimod cream.
* The participant with diagnosis of mild to moderate stable psoriasis vulgaris:
* BSA < 10%.
* PGA ≥ 2.
* Capable of giving written informed consent.

Exclusion Criteria:

* ALT/AST > 3 ULN, BUN/Cr > 1.5 ULN.
* Skin lesions were limited to head，face and skin folds.
* Women who are pregnant, breast-feeding, or planning to become pregnant.
* Known to be allergic to active ingredients or any of the components of the drug.
* Alcoholic, or regular use of Chinese herbs or sedatives, sleeping pills, tranquilizers and other addictive drugs.
* Subjects who have other conditions that may interfere with the evaluation of the efficacy of psoriasis and/or other serious skin diseases other than psoriasis.
* Subjects who have serious diseases of the central nervous system, cardiovascular system, kidney, liver, digestive tract, respiratory system, metabolism and skeletal muscle system.
* Subjects who were considered unsuitable to participate in the study by the investigators.
* Received uv phototherapy, photochemotherapy, or systemic therapy (e.g., systemic glucocorticoid, methotrexate, retinoic acid, or cyclosporine) within 4 weeks prior to baseline visit.
* Received topical anti-psoriasis therapy (including topical glucocorticoids, retinoids, vitamin D analogues, or calcineurin inhibitors) within 2 weeks prior to baseline visit, except where the site of administration was not the target lesion after enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with ≥75% improvement in Psoriasis Area and Severity Index (PASI) score 12 weeks after retreatment with Benvitimod cream or placebo | Week 12
  The PASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema (redness), induration (plaque thickness), and scale, and the extent of %Body Surface Area (BSA) affected with psoriasis. The 3 clinical signs are each graded on a 5-point scale (0 to 4) and the %BSA affected is scored on a 7-point scale (0 to 6) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. Higher scores indicate more severe disease. PASI is a static assessment made without reference to previous scores.

SECONDARY OUTCOMES:
Proportion of participants with ≥90% improvement in Psoriasis Area and Severity Index (PASI) score 12 weeks after retreatment with Benvitimod cream or placebo | Week 12
  The PASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema (redness), induration (plaque thickness), and scale, and the extent of %Body Surface Area (BSA) affected with psoriasis. The 3 clinical signs are each graded on a 5-point scale (0 to 4) and the %BSA affected is scored on a 7-point scale (0 to 6) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. Higher scores indicate more severe disease. PASI is a static assessment made without reference to previous scores.
Proportion of participants who Physician Global Assessment (PGA) score achieved 0 or 1 12 weeks after retreatment with Benvitimod cream or placebo | Week 12
  The PGA is a clinical tool for assessing the current state/severity of a participant's psoriasis at a given timepoint. It is a static 6-point (0-5) morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema, scaling, and plaque thickness/elevation as guidelines. Higher PGA scores represent more severe disease.
Change of Psoriasis Area and Severity Index (PASI) score over time after retreatment with Benvitimod cream or placebo | Week 12
  The PASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema (redness), induration (plaque thickness), and scale, and the extent of %Body Surface Area (BSA) affected with psoriasis. The 3 clinical signs are each graded on a 5-point scale (0 to 4) and the %BSA affected is scored on a 7-point scale (0 to 6) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. Higher scores indicate more severe disease. PASI is a static assessment made without reference to previous scores.
Change of erythema (redness), induration (plaque thickness), and scale score in the skin lesions over time after retreatment with Benvitimod cream or placebo | Week 12
  Change of erythema (redness), induration (plaque thickness), and scale score in the skin lesions over time after retreatment with Benvitimod cream or placebo
Duration of remission after treatment response | Week 12
  Duration of remission after treatment response
The Dermatology Life Quality Index (DLQI) total and individual dimension scores | Week 12
  The DLQI is a simple dermatology-specific 10-question validated questionnaire to assess the impact of the disease on a participant's quality of life. DLQI scores range from 0 to 30, with a higher score indicating a more impaired quality of life.
European Questionnaires Five Dimensions Five Levels (EQ-5D-5L) scores | Week 12
  EQ-5D-5L is a standardized instrument for measuring generic health status. Rated level can be coded as a number 1, 2, 3, 4 or 5, which indicates having no problems for 1, having some problems for 2, having moderate problems for 3, having serious problems for 4 and having extreme problems for 5.
Incidence of AE during the study | Week 16
  AE definition: adverse event
Incidence of SAE during the study | Week 16
  SAE definition: serious adverse event
Incidence of ADR during the study | Week 16
  ADR definition: adverse reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No